CLINICAL TRIAL: NCT02545881
Title: Development and Validation of Novel MRI Methods for the Detection of Prostate Cancer Aggressiveness
Acronym: PROAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Hannu Aronen, Professor, Chief Physician, Turku University Hospital
Other Study IDs: Turku UH
Record Dates: First submitted 2015-08-05; First posted 2015-09-10 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fixed tissue

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — MRI of the prostate prior to prostatectomy

SUMMARY:
The purpose of this study is to develop, validate, and evaluate the correlation of novel magnetic resonance imaging (MRI) methods with prostate cancer aggressiveness and histological data obtained during prostatectomy.

DETAILED DESCRIPTION:
Prostate cancer is one of the most common neoplastic diseases in men. Prostate specific antigen (PSA) has only a limited role in the diagnosis and characterization of prostate cancer. The diagnosis of prostate cancer is still most commonly done by transrectal ultrasonography (TRUS) guided biopsy. However, TRUS guided biopsy carries a risk of increase in complications. There is an increasing interest in developing more accurate non-invasive imaging modalities which could potentially detect prostate cancer aggressiveness.

Diffusion weighted imaging (DWI) and rotating frame relaxation measurements have shown to be particularly promising in prostate cancer detection and characterization. This study which focuses on further development and validation of DWI and rotating frame relaxation measurements will enroll 200 men with histologically diagnosed prostate cancer who will undergo magnetic resonance imaging (MRI) before prostatectomy. Anatomical MRI and novel acquisition methods focusing on DWI and rotating frame relaxation measurements will be performed using surface coils to non-invasively detect and characterize prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35 to 85 years
* Language spoken: Finnish
* Performance status: Karnofsky score 70 or better or WHO performance status 2 or better
* Diagnosis: Histologically confirmed adenocarcinoma of prostate
* No previous surgical, radiation or endocrine treatment for prostate carcinoma
* Clinical stage T1c-T3aN0 based on transrectal ultrasound, pelvic CT and bone scintigraphy
* Time period between the last biopsy and scheduled radical prostatectomy less than 8 months
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* previous prostate surgeries, e.g. TURP (transurethral prostatic resection)
* symptomatic acute prostatitis
* contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* uncontrolled serious infection
* claustrophobia

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically diagnosed prostate cancer who are scheduled for radical prostatectomy in a university hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
MR relaxation values | Within 1 month prior to prostatectomy
  Aim is to study the correlation between MRI parameters (MR relaxation values and different DWI parameters) and histological data including Gleason grade of prostate cancer
MR DWI parameters | Within 1 month prior to prostatectomy
  Aim is to study the correlation between MRI parameters (MR relaxation values and different DWI parameters) and histological data including Gleason grade of prostate cancer
Histological prostate cancer aggressiveness (Gleason grade) | Within 1 month after MR imaging of the prostate
  Aim is to study the correlation between MRI parameters (MR relaxation values and different DWI parameters) and histological data including Gleason grade of prostate cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Turku University Hospital, Turku, Finland